CLINICAL TRIAL: NCT02575638
Title: Phase I Clinical Trial of Camptothecin-20-O-Propionate Hydrate (CZ48)
Brief Title: Safety Study of Camptothecin-20-O-Propionate Hydrate (CZ48)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cao Pharmaceuticals Inc. (Industry)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CZ48-01
Record Dates: First submitted 2015-10-09; First posted 2015-10-15 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Malignant Lymphoma of Extranodal and/or Solid Organ Site; Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment population (Experimental): The study drug, CZ48, is administered orally in capsule form t.i.d. Capsules in 30mg and 50mg of drug are available for dosing. This is a dose escalation study so dosage has not yet been determined. Study drug is take on day 1 - 5 and then no drug on day 6 and 7. This is repeated for 4 weeks, or one course.
  Interventions: Drug: CZ48

INTERVENTIONS:
Drug: CZ48 — CZ48 is an analog of the topoisomerase I inhibitor Camptothecin (CPT). CPT is a natural extract from the tree Camptotheca acuminata
  Other Names: Camptothecin-20-O-Propionate hydrate

SUMMARY:
This is a single-arm, non-randomized feasibility and Phase I trial of 20(S) Camptothecin Propionate administered orally. CZ48 will be administered in successive cohorts of 1 patient per participating site until hints of toxicity (grade 2 or worse adverse events related to the drug) are observed. Then cohorts of 3+3 patients will be treated. CZ48 will be administered orally daily (1 course = 4 weeks). No pre-medications will be administered. Patients will be asked to drink up to one gallon of fluid daily if possible to flush the bladder to mitigate cystitis. Cystitis is an anticipated toxicity as CZ48 is a pro-drug of CPT (Camptothecin)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

• To describe the dose limiting toxicities and adverse event profile of Camptothecin-20-O-Propionate hydrate (CZ48) administered orally every day for 4 weeks (1 course).

SECONDARYOBJECTIVE

* To determine the Maximum Tolerated Dose (MTD) of Camptothecin-20-O-Propionate hydrate (CZ48).
* To determine the blood plasma levels (PK study) of orally administered CZ48.
* To assess responses by Response Evaluation Criteria in Solid Tumors (RECIST) criteria when applicable.
* To follow patients for survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a Performance Status (Zubrod) performance status of 0-1
* Patients must sign an informed consent document
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1,500 /mm3 and platelet count >100,000/mm3 along with an absence of a red blood cell transfusion in the two weeks prior to their participation in the trial
* Patients should have adequate hepatic function with a total bilirubin within normal range and serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) < two times the upper limit of normal (ULN) for patients without liver metastasis and SGOT or SGPT < five times ULN for those with liver metastasis, and adequate renal function as defined by a serum creatinine within 1.5 times the upper limit of normal.
* Patients may receive no other concurrent anticancer treatments such as chemotherapy, hormone therapy (except for prostate cancer patients on luteinizing hormone-releasing hormone ((LHRH)) agonists), immunotherapy, biological agents, investigational agents, or radiation therapy during this trial, and should be off these treatments for at least 2 weeks, or until they have completely recovered from the side effects of these treatments, whichever is longest, except for persistent grade 1 neuropathy in patients who received prior platinum or taxanes.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Patients with brain metastasis that have been treated, asymptomatic and off any steroid use are permitted for study
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception (contraceptive pill, or intrauterine device ((IUD)), or two mechanical barriers).
* Patients with severe uncontrolled medical problems are not eligible for this trial.
* Patients who have too much esterase as determined by a pre-screen dose, with a conversion rate yielding concentration of CPT > 100 ng/ml in vitro.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2008-07; Primary Completion 2019-10-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
To describe the dose limiting toxicities as a measure of the adverse event profile | 4 weeks
  To describe the dose limiting toxicities and adverse event profile of Camptothecin-20-O-Propionate hydrate (CZ48) administered orally for 1 course of treatment.

SECONDARY OUTCOMES:
Determine the Maximum Tolerated Dose (MTD) | 4 weeks
  Using the adverse event profile, the MTD will be established.
Measure the Maximum Concentration (Cmax) level of drug in the blood plasma | 4 weeks
  To measure the blood plasma levels of study drug at various time points to determine Cmax.
Measure the Area Under the Curve (AUC) level of drug in the blood plasma | 4 weeks
  To measure the blood plasma levels of study drug at various time points to determine AUC.
Objective response | 3 months
  To assess responses by RECIST criteria when applicable
Survival | 18 months (measured)
  To follow patients for survival.

CONTACTS AND LOCATIONS:
Overall Officials: Zhisong Cao, Ph. D., Principal Investigator — Cao Pharmaeuticals Inc.
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A study of 9-nitrocamptothecin (RFS-2000) in patients with advanced pancreatic cancer — http://www.ncbi.nlm.nih.gov/pubmed/10200331
- See also: Structure-Activity Relationship of Alkyl 9-Nitrocamptothecin Esters — http://www.chinaphar.com/1671-4083/24/109.htm
- See also: Development and validation of a reverse-phase HPLC (high pressure liquid chromatography) with fluorescence detector method for simultaneous determination of CZ48 and its active metabolite camptothecin in mouse plasma — https://www.infona.pl/resource/bwmeta1.element.elsevier-ded15d2d-7bd7-3a27-890b-e64a8d39932d
- See also: Sulfuric Acid Catalyzed Preparation of Alkyl and Alkenyl Camptothecin Ester Derivatives and Antitumor Activity against Human Xenografts Grown in Nude Mice — http://www.scirp.org/journal/PaperInformation.aspx?PaperID=18169
- See also: Metabolic Difference of CZ48 in Human and Mouse Liver Microsomes — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3382816/
- See also: Antitumor activity of new haloalkyl camptothecin esters against human cancer cell lines and human xenografts grown in nude mice — http://www.ingentaconnect.com/content/ben/acamc/2012/
- See also: Enhanced Lactone Stability of CZ48 in Blood Correlates to its Lack of Toxicity in Mice — http://www.cspsCanada.org